CLINICAL TRIAL: NCT01400581
Title: Collaborative Care for Primary Care Patients With Alcohol Use Disorders
Brief Title: Considering Healthier Drinking Options in Collaborative Care
Acronym: CHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); University of Washington (Other); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01AA018702 (NIH)
Record Dates: First submitted 2011-02-17; First posted 2011-07-22 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collaborative Care [CC] Intervention (Experimental): The CC intervention will consist of offering subjects: 1) an in-depth baseline assessment, 2) frequent (weekly first, then monthly) visits with a nurse care manager, 3) alcohol dependence medications prescribed by a Nurse Practitioner. An interdisciplinary CC team will supervise nurse care managers weekly.
  Interventions: Behavioral: Collaborative Care Intervention
- Usual Care (No Intervention): Observational

INTERVENTIONS:
Behavioral: Collaborative Care Intervention — See description of Intervention arm
  Arms: Collaborative Care [CC] Intervention

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a collaborative care intervention for evidence based management of alcohol use disorders in primary care settings within the Veterans Administration Puget Sound Health Care System (Seattle and American Lake Divisions). The study will test whether patients offered the collaborative care intervention have fewer heavy drinking days at 12 months follow-up and to be abstinent or drinking below recommended limits without problems.

DETAILED DESCRIPTION:
The proposed study will evaluate the effectiveness of a collaborative care intervention for evidence-based management of alcohol use disorders in primary care settings. The investigators will specifically test whether patients offered Collaborative Care:

Have fewer heavy drinking days at 12 months follow-up; and Are more likely to be abstinent or drinking below recommended limits without problems at 12 months follow-up.

Research Design:

The study is a randomized controlled encouragement trial. Consenting patients who complete all baseline assessments will be randomized to be offered the Collaborative Care (CC) intervention or receive Usual Care and will be assessed prospectively. Due to the powerful effect of alcohol assessments on drinking behavior, a cohort of men identified through VISTA/CPRS queries as being potentially eligible for the study will be followed electronically for the following year. A random 25% sample of these men will serve as a "no contact control group" and will have no contact with the study. The remaining 75% will be eligible for screening and recruitment.

Methodology The study will enroll up to 400 subjects (age < 65 years) with probable alcohol use disorders, in order to randomize 300 subjects who complete all baseline assessments. Eligibility criteria include a recent AUDIT-C screening score ≥ 5, phone number available in CPRS, and frequent heavy drinking days in the past four weeks (≥ 5 drinks for men, ≥4 drinks for women).

The CC intervention will consist of offering subjects: 1) an in-depth baseline assessment, 2) frequent (weekly first, then monthly) visits with a nurse care manager, 3) alcohol dependence medications prescribed by a Nurse Practitioner. An interdisciplinary CC team will supervise nurse care managers weekly.

All enrolled participants will have telephone surveys at baseline, 3 months and 12 months; and lab testing at baseline and 12 months. Main study outcomes include: 1) number of heavy drinking days in the past four weeks, and 2) abstinence or drinking below recommended limits at 12 months. Secondary analyses will compare CC and Usual Care groups on process measures of engagement in alcohol-related care, secondary drinking outcomes, laboratory markers, health-related quality of life, health care utilization, and health care costs. For the observational cohort, secondary analyses will compare drinking behaviors (AUDIT-C scores), alcohol-related diagnoses, and health care utilization between men who have no contact with study procedures and other subgroups who are eligible for screening and recruitment.

The investigators hypothesize that subjects in the intervention group will decrease their frequency of heavy drinking and will be more likely to be abstinent or drinking below recommended limits at 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* AUDIT-C score 5 or more (modification described below)
* Age less than 65 at time of AUDIT-C screen (modification described below)
* Phone number available in electronic medical record
* Frequent heavy drinking reported during brief telephone screen (8 heavy drinking days in past 4 weeks, 5 or more drinks in a day for men, 4 or more for women; OR 4 heavy drinking days past four weeks and prior alcohol treatment or attendance at AA)

Exclusion Criteria:

* Missing address or phone number in electronic medical record
* Warning flag regarding violent behavior in medical record
* Patient participating in addictions treatment
* Primary care provider or patient indicates not to contact patient
* Barriers to telephone assessment (hearing, non-English)
* Unable to provide adequate collateral contacts
* Cognitive impairment
* Unstable or acute medical, surgical, or psychiatric problem requiring emergency care
* Not available for follow-up (planning to move, life expectancy <1 yr, hospice)
* Pregnancy
* VA employee

Prior to the start of the trial these changes were made (VA IRB approval: 8/2011):

* Changed from AUDIT-C score ≥5 for both men and women TO: AUDIT-C score ≥5 for men; AUDIT-C score ≥4 for women (to increase the pool of potentially eligible women)
* From age 65 years and younger to age ≤75 years

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 304 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
1) number of heavy drinking days | at 12 months
2) abstinence or drinking below recommended limits without problems | at 12 months

SECONDARY OUTCOMES:
Engagement in alcohol-related care | 12-months
secondary drinking outcomes and laboratory markers | 12-months
health-related quality of life | 12-months
health care utilization | 12-months
health care costs | 12-months
Outcomes 1-7 listed above and secondary drinking, readiness to change, and engagement outcomes. | at 3-months

CONTACTS AND LOCATIONS:
Overall Officials: Katharine A Bradley, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Background] Bradley KA, Ludman EJ, Chavez LJ, Bobb JF, Ruedebusch SJ, Achtmeyer CE, Merrill JO, Saxon AJ, Caldeiro RM, Greenberg DM, Lee AK, Richards JE, Thomas RM, Matson TE, Williams EC, Hawkins E, Lapham G, Kivlahan DR. Patient-centered primary care for adults at high risk for AUDs: the Choosing Healthier Drinking Options In primary CarE (CHOICE) trial. Addict Sci Clin Pract. 2017 May 17;12(1):15. doi: 10.1186/s13722-017-0080-2. PMID 28514963
- [Result] Bradley KA, Bobb JF, Ludman EJ, Chavez LJ, Saxon AJ, Merrill JO, Williams EC, Hawkins EJ, Caldeiro RM, Achtmeyer CE, Greenberg DM, Lapham GT, Richards JE, Lee AK, Kivlahan DR. Alcohol-Related Nurse Care Management in Primary Care: A Randomized Clinical Trial. JAMA Intern Med. 2018 May 1;178(5):613-621. doi: 10.1001/jamainternmed.2018.0388. PMID 29582088
- [Derived] Williams EC, Bobb JF, Lee AK, Ludman EJ, Richards JE, Hawkins EJ, Merrill JO, Saxon AJ, Lapham GT, Matson TE, Chavez LJ, Caldeiro R, Greenberg DM, Kivlahan DR, Bradley KA. Effect of a Care Management Intervention on 12-Month Drinking Outcomes Among Patients With and Without DSM-IV Alcohol Dependence at Baseline. J Gen Intern Med. 2019 Dec 10. doi: 10.1007/s11606-019-05261-7. Online ahead of print. PMID 31432438
- [Derived] Takahashi T, Lapham G, Chavez LJ, Lee AK, Williams EC, Richards JE, Greenberg D, Rubinsky A, Berger D, Hawkins EJ, Merrill JO, Bradley KA. Comparison of DSM-IV and DSM-5 criteria for alcohol use disorders in VA primary care patients with frequent heavy drinking enrolled in a trial. Addict Sci Clin Pract. 2017 Jul 18;12(1):17. doi: 10.1186/s13722-017-0082-0. PMID 28716049

DOCUMENTS (1):
  • Informed Consent Form (2012-03-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT01400581/ICF_000.pdf